CLINICAL TRIAL: NCT02014428
Title: Oral Low-molecular Weight Hyaluronic Acid in the Treatment of Atrophic Vaginitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: HA-123
Record Dates: First submitted 2013-12-09; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Hyaluronic Acid

ARMS (2):
- Hyaluronic acid (Experimental): 220 mg hyaluronic acid per tablet (two tablets/day for 10 days, and subsequently one tablet/day for three months)
  Interventions: Dietary Supplement: Hyaluronic acid
- Placebo (Placebo Comparator): two tablets/day for 10 days, and subsequently one tablet/day for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Hyaluronic acid
  Arms: Hyaluronic acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of low molecular weight hyaluronic acid oral tablets for the treatment of atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* at least 12 months postmenopausal
* mucosal atrophy and the main bothersome related symptoms, such as itching, burning, and dyspareunia.

Ages: 45 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Atrophic vaginal changes | Change from baseline epithelium at 3 months
  Morphometric analysis of biopsies.

SECONDARY OUTCOMES:
Assessment of Itching | Change from baseline Itching at 3 months
  Scale: absent, mild, moderate, severe.
Assessment of Burning | Change from baseline Burning at 3 months
  Scale: absent, mild, moderate, severe.
Assessment of Dyspareunia | Change from baseline Dyspareunia at 3 months
  Scale: absent, mild, moderate, severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecological, Obstetric Sciences and Reproductive Medicine, University of Messina., Messina, Italy